CLINICAL TRIAL: NCT03753087
Title: A Phase 4, Single-center, Randomized, Parallel Group Study to Assess Effects of Empagliflozin on Exercise Capacity and Left Ventricular Diastolic Function in Patients With Heart Failure With Preserved Ejection Fraction and Type-2 Diabetes Mellitus
Brief Title: Effects of Empagliflozin on Exercise Capacity and Left Ventricular Diastolic Function in Patients With Heart Failure With Preserved Ejection Fraction and Type-2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Collaborators: Ministry of Health, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Anton Borisov, Principal Investigator, MD, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-9-25
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure, Diastolic; Diabetes Mellitus, Type 2
Keywords: HF; HFpEF; DM; Empagliflozin; Jardiance
MeSH Terms: conditions — Heart Failure, Diastolic; Diabetes Mellitus, Type 2 | interventions — empagliflozin; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Patients will receive standard care for Heart Failure and Diabetes Mellitus + Empagliflozin 10mg once daily
  Interventions: Drug: Empagliflozin
- Control (Active Comparator): Patients will receive standard care for Heart Failure and Diabetes Mellitus with no SGLT-2 inhibitors
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Empagliflozin — 10 mg tablet
  Arms: Empagliflozin
Other: Standard care — Standard care with no SGLT-2 inhibitors
  Arms: Control

SUMMARY:
Patients enrolled into the study will be randomly allocated either to Empagliflozin group or control group. In the Empagliflozin group patients will be receiving standard care + Empagliflozin 10 mg o.d., in the control group patients will be receiving standard care without sodium glucose contransporter 2 (SGLT2) inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 45 to 80 years at screening
2. Diagnosis of type-2 diabetes mellitus with stable glucose-lowering background therapy for at least 12 weeks
3. HbA1c ≥ 6,5% and ≤ 10% at screening
4. Diagnosis of HFpEF which includes:

   * Symptoms ± signs (as defined in 2016 European Society of Cardiology guidelines for the diagnosis and treatment of acute and chronic heart failure)
   * Ejection fraction ≥ 50% (by Simpson)
   * Increased LV filling pressures at rest or during exercise determined by echocardiography (LV diastolic dysfunction grade II/III and/or positive diastolic stress test) [according to American Society of Echocardiography and European Association of Cardiovascular Imaging (ASE/EACVI) Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography, 2016]
5. Signed and dated informed consent

Exclusion Criteria:

1. Pretreatment with empagliflozin or other SGLT-2 inhibitor within the last 2 months
2. Type-1 diabetes mellitus
3. NYHA classification IV or acute decompensated heart failure at screening
4. Impaired renal function, defined as eGFR <30 ml/min/1.73 m² of body-surface-area (CKD-EPI)
5. Systolic blood pressure > 180 mmHg or < 90 mmHg
6. Permanent atrial flutter or atrial fibrillation
7. Other conditions that may be responsible for impaired diastolic function such as hypertrophic/restrictive cardiomyopathy, constrictive pericarditis and etc.
8. Anemia (Hb < 100 g/l)
9. Myocardial infarction, coronary artery bypass graft surgery within the last 3 months
10. Stroke or TIA within the last 3 months
11. Indications of liver disease
12. Acute genital infection or urinary tract infection
13. Pregnancy
14. Additional exclusion criteria may apply

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walking distance (6MWD) | 24 weeks
  Difference in distance walked during 6-minute walking test (6MWT) between 24 weeks after baseline and at baseline

SECONDARY OUTCOMES:
Change in left ventricular mass index (LVMI) | 24 weeks
  Difference in LVMI assessed by echocardiography between 24 weeks after baseline and at baseline
Change in left atrial volume index (LAVI) | 24 weeks
  Difference in LAVI assessed by echocardiography between 24 weeks after baseline and at baseline
Change in left atrial stiffness | 24 weeks
  Difference in left atrial stiffness assessed as a ratio of mitral E/e' ratio to left atrial strain s between 24 weeks after baseline and at baseline
Change estimated pulmonary artery systolic pressure (PASP) | 24 weeks
  Difference in PASP assessed by echocardiography both at rest and during diastolic stress test (DST) between 24 weeks after baseline and at baseline
Change in average e' velocity | 24 weeks
  Difference in average e' velocity assessed by echocardiography both at rest and during diastolic stress test (DST) between 24 weeks after baseline and at baseline
Change in average E/e' ratio | 24 weeks
  Difference in average E/e' ratio assessed by echocardiography both at rest and during diastolic stress between 24 weeks after baseline and at baseline
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) | 24 weeks
  Difference in NT-proBNP plasma levels between 24 weeks after baseline and at baseline
Change in Cyclic guanosine monophosphate (cGMP) | 24 weeks
  Difference in cGMP plasma levels between 24 weeks after baseline and at baseline
Change in Endothelin 1 (ET-1) | 24 weeks
  Difference in ET-1 plasma levels between 24 weeks after baseline and at baseline
Change in Growth/differentiation factor 15 (GDF-15) | 24 weeks
  Difference in GDF-15 plasma levels between 24 weeks after baseline and at baseline
Change in ST2 | 24 weeks
  Difference in ST2 plasma levels between 24 weeks after baseline and at baseline
Change in Galectin-3 | 24 weeks
  Difference in Galectin-3 plasma levels between 24 weeks after baseline and at baseline
Change in carboxyterminal propeptide of type I collagen (PICP) | 24 weeks
  Difference in PICP plasma levels between 24 weeks after baseline and at baseline
Change in Human Pentraxin 3 (PTX3) | 24 weeks
  Difference in PTX3 plasma levels between 24 weeks after baseline and at baseline
Change in high-sensitivity C-reactive protein (hsCRP) | 24 weeks
  Difference in hsCRP plasma levels between 24 weeks after baseline and at baseline
Change in Interleukin-6 (IL-6) | 24 weeks
  Difference in IL-6 plasma levels between 24 weeks after baseline and at baseline
Change of New York Heart Association (NYHA) functional classification | 24 weeks
  Difference in NYHA class between 24 weeks after baseline and at baseline
Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) score | 24 weeks
  Difference in MLHFQ score between 24 weeks after baseline and at baseline.
  The questionnaire is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses.
  Score ranges from 0 (best quality of life) to 105 (worst quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Anton Borisov, MD, Principal Investigator — National Medical Research Center for Cardiology
Locations (1):
- National Medical Research Center for Cardiology, Moscow, Russia

REFERENCES:
- [Derived] Ovchinnikov A, Potekhina A, Filatova A, Svirida O, Zherebchikova K, Ageev F, Belyavskiy E. Effects of empagliflozin on functional capacity, LV filling pressure, and cardiac reserves in patients with type 2 diabetes mellitus and heart failure with preserved ejection fraction: a randomized controlled open-label trial. Cardiovasc Diabetol. 2025 May 9;24(1):196. doi: 10.1186/s12933-025-02756-y. PMID 40346546